CLINICAL TRIAL: NCT00269672
Title: A Randomized, Open Label, Controlled Phase II Study to Evaluate Safety, Tolerability and Immunogenicity After Two Different 13-Valent Pneumococcal Conjugate Vaccine Formulations in Elderly Subjects Aged 65 Years and Older Who Are Naive to Previous 23vPS Immunization
Brief Title: Study to Evaluate a 13-valent Pneumococcal Conjugate Vaccine in Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6115A1-500
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2010-08

CONDITIONS: Vaccines, Pneumococcal Conjugate Vaccine
Keywords: vaccine

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine

SUMMARY:
There is evidence that aluminum phosphate (AlPO4) contained as an adjuvant in conjugate vaccines enhances the immune response in infants. There is no data so far evaluating whether this also applies to adults. The objective of this study is to compare the immune response of 2 different 13-valent pneumococcal conjugate (13vPnC) formulations with and without AlPO4 to select a formulation and to compare the immune response to the chosen 13vPnC formulation relative to the immune response to 23-valent pneumococcal polysaccharide vaccine (23vPS).

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults 65 years of age and older.
* Determined by medical history, physical examination, and clinical judgment to be eligible for the study.
* Expected to be available for the duration of the trial (up to approximately 13 months).

Exclusion Criteria:

* Received previous immunization with 23vPS.
* Serious chronic disorders including metastatic malignancy
* Known or suspected hypersensitivity to any vaccine or vaccine components

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 915 (Actual)
Dates: Start 2005-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Demonstrate 13vPnC without AlPO4 is as immunogenic as 13vPnC with AlPO4 to select a 13vPnC formulation.

SECONDARY OUTCOMES:
Demonstrate that the selected 13vPnC formulation is as immunogenic as 23vPS (by IgG).
Safety and tolerability of the selected 13vPnC formulation given 12 months after a previous dose of the selected 13vPnC.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Juergens C, de Villiers PJ, Moodley K, Jayawardene D, Jansen KU, Scott DA, Emini EA, Gruber WC, Schmoele-Thoma B. Safety and immunogenicity of 13-valent pneumococcal conjugate vaccine formulations with and without aluminum phosphate and comparison of the formulation of choice with 23-valent pneumococcal polysaccharide vaccine in elderly adults: a randomized open-label trial. Hum Vaccin Immunother. 2014;10(5):1343-53. doi: 10.4161/hv.27998. Epub 2014 Feb 27. PMID 24576885